CLINICAL TRIAL: NCT03694418
Title: We Are Here Now: a Multi-level, Multicomponent Sexual and Reproductive Health Intervention for American Indian Youth
Acronym: NE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: Northern Arizona University (Other); Fort Peck Community College (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Elizabeth Rink, Professor, Montana State University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: R01MD012761 (NIH); R01MD012761 (NIH)
Record Dates: First submitted 2018-09-28; First posted 2018-10-03 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Reproductive Behavior; Sexual Behavior
MeSH Terms: conditions — Reproductive Behavior; Sexual Behavior

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cluster 1 (Other): Cluster 1 is 1 school on the Fort Peck Reservation that will be randomized into the intervention in 2019. Cluster 1 will receive all four levels of the intervention including: 1) A school-based SRH curriculum called Native Stand, designed to address individual-level factors that lead to sexual risk behaviors; 2) a family-level curriculum called Native Voices, tailored to increase communication between adult family members and youth about SRH topics; 3) a cultural mentoring component at the community level that pairs AI youth with adults and elders to discuss traditional AI beliefs and practices about SRH; and 4) a mobilizing strategy to activate a multi-sectoral network of youth-servicing organizations at the systems level in Fort Peck to coordinate SRH services for AI youth.
  Interventions: Behavioral: We are here now: a multi-level, multi-component sexual and reproductive health intervention for American Indian youth
- Cluster 2 (Other): Cluster 2 includes 1 school on the Fort Peck Reservation that will be randomized in the intervention in 2019-2020. Cluster 2 will receive all four levels of the intervention including: 1) A school-based SRH curriculum called Native Stand, designed to address individual-level factors that lead to sexual risk behaviors; 2) a family-level curriculum called Native Voices, tailored to increase communication between adult family members and youth about SRH topics; 3) a cultural mentoring component at the community level that pairs AI youth with adults and elders to discuss traditional AI beliefs and practices about SRH; and 4) a mobilizing strategy to activate a multi-sectoral network of youth-servicing organizations at the systems level in Fort Peck to coordinate SRH services for AI youth.
  Interventions: Behavioral: We are here now: a multi-level, multi-component sexual and reproductive health intervention for American Indian youth
- Cluster 3 (Other): Cluster 3 includes 1 school on the Fort Peck reservation that will be randomized into the intervention in 2020-2021. Cluster 3 will receive all four levels of the intervention including: 1) A school-based SRH curriculum called Native Stand, designed to address individual-level factors that lead to sexual risk behaviors; 2) a family-level curriculum called Native Voices, tailored to increase communication between adult family members and youth about SRH topics; 3) a cultural mentoring component at the community level that pairs AI youth with adults and elders to discuss traditional AI beliefs and practices about SRH; and 4) a mobilizing strategy to activate a multi-sectoral network of youth-servicing organizations at the systems level in Fort Peck to coordinate SRH services for AI youth.
  Interventions: Behavioral: We are here now: a multi-level, multi-component sexual and reproductive health intervention for American Indian youth
- Cluster 4 (Other): Cluster 4 includes 1 school on the Fort Peck reservation that will be randomized into the intervention in 2020-2021. Cluster 4 will receive all four levels of the intervention including: 1) A school-based SRH curriculum called Native Stand, designed to address individual-level factors that lead to sexual risk behaviors; 2) a family-level curriculum called Native Voices, tailored to increase communication between adult family members and youth about SRH topics; 3) a cultural mentoring component at the community level that pairs AI youth with adults and elders to discuss traditional AI beliefs and practices about SRH; and 4) a mobilizing strategy to activate a multi-sectoral network of youth-servicing organizations at the systems level in Fort Peck to coordinate SRH services for AI youth.
  Interventions: Behavioral: We are here now: a multi-level, multi-component sexual and reproductive health intervention for American Indian youth
- Cluster 5 (Other): Cluster 5 includes 1 school on the Fort Peck reservation that will be randomized into the intervention in 2020-2021. Cluster 4 will receive all four levels of the intervention including: 1) A school-based SRH curriculum called Native Stand, designed to address individual-level factors that lead to sexual risk behaviors; 2) a family-level curriculum called Native Voices, tailored to increase communication between adult family members and youth about SRH topics; 3) a cultural mentoring component at the community level that pairs AI youth with adults and elders to discuss traditional AI beliefs and practices about SRH; and 4) a mobilizing strategy to activate a multi-sectoral network of youth-servicing organizations at the systems level in Fort Peck to coordinate SRH services for AI youth.
  Interventions: Behavioral: We are here now: a multi-level, multi-component sexual and reproductive health intervention for American Indian youth

INTERVENTIONS:
Behavioral: We are here now: a multi-level, multi-component sexual and reproductive health intervention for American Indian youth — N/E will be implemented simultaneously over the 9-month school year. Components include: 1) Individual Level- Native Stand 2) Family Level - Native Voices; 3) Community Level - Cultural mentoring program; and 4) Systems Level. The fourth level of N/E mobilizes the existing Epidemiology Team to enhance the coordination and implementation of SRH services at Fort Peck.

SUMMARY:
N/E is a community-based participatory research (CBPR) multi-level, multi-component sexual and reproductive health (SRH) intervention, constructed on Ecological Systems Theory. N/E is based on Fort Peck tribal members' desire to implement a holistic SRH intervention for American Indian youth. N/E includes: 1) A school-based SRH curriculum called Native Stand, designed to address individual-level factors that lead to sexual risk behaviors; 2) a family-level curriculum called Native Voices, tailored to increase communication between adult family members and youth about SRH topics; 3) a cultural mentoring component at the community level that pairs American Indian youth with adults and elders to discuss traditional American Indian beliefs and practices about SRH; and 4) a mobilizing strategy to activate a multi-sectoral network of youth-servicing organizations at the systems level in Fort Peck to coordinate SRH services for American Indian youth. The overarching aim of this proposal is to refine, tailor, and finalize the components of N/E and evaluate its efficacy. We will use a cluster-randomized stepped-wedge design (SWD), in which 5 schools that American Indian youth from Fort Peck attend are the clusters to be randomized into the intervention 1 at a time, with all schools eventually being randomized to the intervention. The 5 schools are located in separate communities, mitigating the potential for cross-contamination. N/E is a 5-year study involving 456 14- to 18-year-old American Indian youth.

DETAILED DESCRIPTION:
N/E is a community-based participatory research (CBPR) multi-level, multi-component sexual and reproductive health (SRH) intervention, constructed on Ecological Systems Theory. N/E is based on Fort Peck tribal members' desire to implement a holistic SRH intervention for American Indian youth. N/E includes: 1) A school-based SRH curriculum called Native Stand, designed to address individual-level factors that lead to sexual risk behaviors; 2) a family-level curriculum called Native Voices, tailored to increase communication between adult family members and youth about SRH topics; 3) a cultural mentoring component at the community level that pairs American Indian youth with adults and elders to discuss traditional American Indian beliefs and practices about SRH; and 4) a mobilizing strategy to activate a multi-sectoral network of youth-servicing organizations at the systems level in Fort Peck to coordinate SRH services for American Indian youth. The overarching aim of this proposal is to refine, tailor, and finalize the components of N/E and evaluate its efficacy. We will use a cluster-randomized stepped-wedge design (SWD), in which 5 schools that American Indian youth from Fort Peck attend are the clusters to be randomized into the intervention 1 at a time, with all schools eventually being randomized to the intervention. The 5 schools are located in separate communities, mitigating the potential for cross-contamination. N/E is a 5-year study involving 456 14- to 18-year-old American Indian youth.

Our specific aims are:

AIM 1: Refine, tailor, and finalize the components of N/E. Our community advisory board and the Fort Peck-based and MSU-based research team will design culturally appropriate adaptations for N/E's 4 levels during the first year of the study, based on the analysis of our recently completed qualitative and quantitative research (focus groups, interviews, and surveys), as well as discussions with elders and community stakeholders.

AIM 2: Test the efficacy of N/E for 14- to 18-year-old American Indian youth. Our hypotheses are:

H1: American Indian youth who participate in N/E will demonstrate increased condom use at 3, 9, and 12 months. (12 months will be used in the Primary Outcome analysis; 3 and 9 months will be used in the Secondary Outcomes analysis.) H2: American Indian youth who participate in N/E will demonstrate increased use of other birth control at 3, 9, and 12 months. They also will demonstrate a decrease in sexual risk behaviors as measured by reduced number of sex partners, delayed onset of sexual intercourse, and decreased substance use during sex, at 3, 9, and 12 months. (Secondary Outcomes) H3: N/E parents/legal guardians and youth will demonstrate significantly increased communication about topics related to SRH at 3, 9, and 12 months. American Indian youth who participate in the cultural mentoring program will demonstrate significantly increased understanding of cultural values related to traditional American Indian beliefs regarding SRH at 3, 9, and 12 months. And American Indian youth who participate in N/E will report significantly increased use of SRH services at 3, 9, and 12 months as a result of improved coordination among education, health care, and social service agencies on the Fort Peck Reservation. (Tertiary Outcomes) AIM 3: Evaluate the fidelity and acceptability of N/E. N/E's fidelity and acceptability will be evaluated using qualitative methods, including focus groups, activity logs, and staff field notes and meetings.

ELIGIBILITY:
Inclusion Criteria:

* 14 to 18 years old
* a registered member of a federally recognized tribe or an associate tribal member
* a resident of Fort Peck with a parent/legal guardian. Exclusion criteria are minimal due to the CAB's value of inclusion in the intervention.
* For inclusion in the systems-level component of the intervention, only those staff members who sit on the Epi Team as representatives of their respective agencies are eligible.

Exclusion Criteria:

* not meeting the aforementioned inclusion criteria
* having a medically identified physical or cognitive impairment that would impede their understanding of and participation in the educational content and activities of Native Stand, Native Voices, and the cultural mentoring program.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 453 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth L Rink, PhD, Principal Investigator — Montana State University
Locations (2):
- United States (2):
  - Montana State University, Bozeman, Montana
  - Fort PeckCommunity College, Poplar, Montana

IPD SHARING:
Plan to Share IPD: No
There is no plan to have an IPD sharing plan at this point in time.

REFERENCES:
- [Derived] Anastario M, Rink E, Firemoon P, Carnegie N, Johnson O, Peterson M, Rodriguez AM. Evidence of secular trends during the COVID-19 pandemic in a stepped wedge cluster randomized trial examining sexual and reproductive health outcomes among Indigenous youth. Trials. 2023 Apr 1;24(1):248. doi: 10.1186/s13063-023-07223-1. PMID 37004106
- [Derived] Rink E, Anastario M, Peterson M, FireMoon P, Johnson O, GrowingThunder R, Ricker A, Cox G, Holder S, Baldwin JA. Baseline results from NenUnkUmbi/EdaHiYedo: A randomized clinical trial to improve sexual and reproductive health among American Indian adolescents. J Adolesc. 2023 Jun;95(4):844-859. doi: 10.1002/jad.12158. Epub 2023 Mar 8. PMID 36890753
- [Derived] Rink E, Firemoon P, Anastario M, Johnson O, GrowingThunder R, Ricker A, Peterson M, Baldwin J. Rationale, Design, and Methods for Nen Unkumbi/Edahiyedo ("We Are Here Now"): A Multi-Level Randomized Controlled Trial to Improve Sexual and Reproductive Health Outcomes in a Northern Plains American Indian Reservation Community. Front Public Health. 2022 Jul 13;10:823228. doi: 10.3389/fpubh.2022.823228. eCollection 2022. PMID 35910931
- [Derived] Rink E, Knight K, Ellis C, McCormick A, FireMoon P, Held S, Webber E, Adams A. Using Community-Based Participatory Research to Design, Conduct, and Evaluate Randomized Controlled Trials with American Indian Communities. Prev Chronic Dis. 2020 Nov 12;17:E143. doi: 10.5888/pcd17.200099. PMID 33180688

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from January 2019 to May 2019. Recruitment included meetings with tribal and school leadership and letters to caregivers who had a child 14- to 18 years old and was attending school.
Groups:
- Cluster 1: Baseline, Then 12 Months NE Intervention: Cluster 1 was implemented from September 2019 to September 2020. The Cluster 1 NE intervention took place from September 2019 to March 2020. The NE intervention was severely impacted by the COVID-19 pandemic and not implemented from March 2020 to May 2020. 12 month data was collected in September 2020.
- Cluster 2: 12 Months Baseline, Then 12 Months NE Intervention: Cluster 2 was implemented from January 2021 to September 2021. Cluster 2 started 4 months later than planned due to the COVID-19 pandemic and the school being closed. In Cluster 2 the NE intervention was implemented from January 2021 to May 2021. 12 month data collection took place in September 2021. Although Cluster 2 had a late start date the intervention was completed as planned.
- Cluster 3: 24 Months Baseline, Then 12 Months NE Intervention: Cluster 3 was implemented from September 2021 to September 2022. The NE intervention in Cluster 3 was implemented from September 2021 to May 2022. 12 month data collection was completed in September 2022.
- Cluster 4: 24 Months Baseline, Then 12 Months NE Intervention: Cluster 4 was implemented from September 2021 to September 2022. Cluster 4 was implemented simultaneously with Cluster 3. The NE intervention was implemented from September 2021 to May 2022, at the same time as Cluster 3. 12 month collection was completed in September 2022.
- Cluster 5: 36 Months Baseline, Then 12 Months NE Intervention: Cluster 5 was implemented from September 2022 to September 2023. The NE intervention was implemented from September 2022 to May 2023. 12 month data collection was completed in September 2023.
Period: Overall Study
Arm/Group | Cluster 1: Baseline, Then 12 Months NE Intervention | Cluster 2: 12 Months Baseline, Then 12 Months NE Intervention | Cluster 3: 24 Months Baseline, Then 12 Months NE Intervention | Cluster 4: 24 Months Baseline, Then 12 Months NE Intervention | Cluster 5: 36 Months Baseline, Then 12 Months NE Intervention
Started | 210 (Cluster 1 took place from September 2019 to September 2020. Cluster 1 impacted by the COVID-19 pandemic during Montana shelter in place orders March 2020 to May 2020. Intervention delivery was not completed from March 2020 to May 2020. The 12 month data collection took place in September 2020.) | 41 (The implementation of Cluster 2 was truncated by the COVID 19 pandemic due to repeated outbreaks occurring in Cluster 2. As a result, Cluster 2 NE intervention delivery took place between January 2021 to May 2021. 24 month data collection took place in September 2021.) | 23 (Cluster 3 was implemented from September 2021 to September 2022 and implemented simultaneously with Cluster 4. The NE intervention was implemented from September 2021 to May 2022. 36 month data collection was completed in September 2022 for Cluster 3.) | 29 (Cluster 4 took place from September 2021 to September 2022 and was implemented simultaneously with Cluster 3. The NE intervention in Cluster 4 took place from September 2021 to May 2022. 36 month data collection in Cluster 4 took place in September 2022.) | 150 (Cluster 5 was implemented from September 2022 to September 2023. The NE intervention in Cluster 5 was implmented from September 2022 to May 2023. The 60 month data collection was completed in September 2023.)
Completed | 95 | 18 | 11 | 17 | 137
Not Completed | 115 | 23 | 12 | 12 | 13
Not completed — Lost to Follow-up | 115 | 23 | 12 | 12 | 13

BASELINE CHARACTERISTICS:
Population: Participants contributed behavioral data on variables related to sexual risk taking.
Groups:
- Cluster 1: Cluster 1 took place from September 2019 to September 2020. Baseline, mid-intervention, and 3 month post intervention data was collected. The Covid-19 pandemic prevented the collection of of the post intervention data.
- Cluster 2: Cluster 2 took place from January 2021 to September 2021. Baseline, mid-intervention, post-intervention, and 3 month post intervention were collected. However, data collection was truncated due to the school in cluster 2 being closed because of the COVID-19 pandemic. Data was collected from January 2021 to September 2021.
- Cluster 3: Cluster 3 took place from September 2021 to September 2022. Baseline, mid-intervention, post-intervention, and 3 month post intervention were collected as planned.
- Cluster 4: Cluster 4 took place from September 2021 to September 2022 simultaneously with Cluster 3. Baseline, mid-intervention, post-intervention, and 3 month post intervention were collected as planned.
- Cluster 5: Cluster 5 took place from September 2022 to September 2023. Baseline, mid-intervention, post-intervention, and 3 month post intervention were collected as planned.
- Total: Total of all reporting groups
Arm/Group | Cluster 1 | Cluster 2 | Cluster 3 | Cluster 4 | Cluster 5 | Total
Number analyzed (Participants) | 210 | 41 | 23 | 29 | 150 | 453
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.7 (1.5) | 15.9 (1.8) | 15.5 (1.4) | 15.0 (1.5) | 15.6 (1.4) | 15.6 (1.5)
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.7 (1.5) | 15.9 (1.8) | 15.5 (1.4) | 15.0 (1.5) | 15.6 (1.4) | 15.6 (1.5)
Age, Customized [Mean (Standard Deviation); unit: years]
  Age of participants | 15.7 (1.5) | 15.9 (1.8) | 15.5 (1.4) | 15.0 (1.5) | 15.6 (1.4) | 15.5 (1.5)
Sex/Gender, Customized [Number; unit: participants] — Gender was measured as a binary variable 1 = male, 0 = female.
  participants
    Student gender (number that are male) by cluster. | 107 | 14 | 9 | 13 | 82 | 225
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 28 | 14 | 16 | 68 | 229
  Male | 107 | 13 | 9 | 13 | 82 | 224
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Participants in study are American Indian.
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 210 | 41 | 23 | 29 | 150 | 453
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 210 | 41 | 23 | 29 | 150 | 453
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 210 | 41 | 23 | 29 | 150 | 453
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 210 | 41 | 23 | 29 | 150 | 453
Number of protected anal or vaginal intercourse acts in past 30 days [Mean (Full Range); unit: proportion of protected sex acts] | 0.40 [0.26 to 0.54] | 0.40 [0.26 to 0.54] | 0.40 [0.26 to 0.54] | 0.40 [0.26 to 0.54] | 0.40 [0.26 to 0.54] | 0.40 [0.26 to 0.54]

OUTCOME MEASURES:

1. Primary Outcome: Number of Protected Acts of Vaginal and/or Anal Sex in the Past 30 Days.
Description: Number of protected acts of sex using a condom during vaginal and/or anal sex in the past 30 days is measured as proportion of condom use during vaginal/anal sex using 2 items (number of times condom used relative to number of times had vaginal/anal sex).
Time Frame: Measure for within the past 30 days from completing survey at 3 months, 9 months, 12 months; data at 12 months reported.
Population: American Indian youth ages 14 - 18 years who are enrolled in a federally recognized tribe and living on the Fort Peck Reservation in Montana.
Measure: Mean (95% Confidence Interval); unit: proportion
Groups:
- NE Intervention: Primary outcome measure is reported for all clusters during the intervention period and was assessed for changes from baseline to 3 month post intervention.
Arm/Group | NE Intervention
Number analyzed (Participants) | 453
proportion | 0.31 [0.15 to 0.47]
Statistical Analysis 1: Comparison: NE Intervention; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney); Incident Rate Ratio = 1.73, 95% CI 2-sided [1.02 to 2.95], Standard Deviation 0.35

2. Secondary Outcome: Ever Had Vaginal and/or Sexual Intercourse.
Description: Measured as a binary yes/no variable. 1 = yes, 0 = no.
Time Frame: Measured at time of survey
Reporting Status: Not Posted, anticipated posting 2025-09

3. Secondary Outcome: Number of Sex Partners in the Past 30 Days.
Description: Number of sex partners in the past 30 days is measured as an integer with no upper limit.
Time Frame: Measured at time of survey completion.
Reporting Status: Not Posted, anticipated posting 2025-09

4. Secondary Outcome: Frequency of Vaginal and/or Anal Sex in the Past 30 Days.
Description: Frequency of vaginal and/or anal sex in the past 30 days is measured as an integer with no upper limit.
Time Frame: Time frame is assessed as within the past 30 days from survey completion.
Reporting Status: Not Posted, anticipated posting 2025-09

5. Secondary Outcome: Change in Number of Pregnancies at 3 Months, 9 Months and 12 Months
Description: Change in number of pregnancies will be measure with 1 item (number of pregnancies)
Time Frame: 3 months, 9 months and 12 months
Reporting Status: Not Posted, anticipated posting 2025-09

6. Secondary Outcome: Frequency of Birth Control Use.
Description: Number of times used birth control during vaginal sex.
Time Frame: Time frame is measured as the past year.
Reporting Status: Not Posted, anticipated posting 2025-09

7. Secondary Outcome: Substance Use During Sex.
Description: Substance use during sex is measured as a binary variable 1 = yes, 0 = no.
Time Frame: Time frame is the past 30 days.
Reporting Status: Not Posted, anticipated posting 2025-09

8. Other Pre Specified Outcome: Change in Increased Parent/Legal Guardian-child Communication About Sexual and Reproductive Health Topics at 3 Months, 9 Months and 12 Months
Description: Change in increased parent/legal-child communication about sexual and reproductive health topics will be measured using a 24 item Likert scale, higher score = higher communication
Time Frame: 3 months, 9 months and 12 months
Reporting Status: Not Posted, anticipated posting 2025-09

9. Other Pre Specified Outcome: Change in Increased Usage of Sexual and Reproductive Health Services at 3 Months, 9 Months and 12 Months
Description: Change in increased usage of sexual and reproductive health services will be measured with 9 items ( frequency, type and follow up of sexual and reproductive health services used)
Time Frame: 3 months, 9 months and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at baseline, 3 months, 9 months, and 12 months for participants in NE. Cluster 1 adverse events were assessed September 2019-September 2020; Cluster 2 adverse events were assessed September 2020-September 2021; Cluster 3 & Cluster 4 adverse events were assessed September 2021-September 2022; Cluster 5 adverse events were assessed September 2022-September 2023. No adverse events were reported during NE.
Description: There were approximately 453 participants at risk for serious adverse events and all-cause mortality.
Groups:
- Cluster 1: Cluster 1 adverse event data was collected over a 12 month period between September 2019 - September 2020.
- Cluster 2: Cluster 2 adverse event data was collected over a 12 month period between September 2020 - September 2021.
- Cluster 3: Cluster 3 adverse event data was collected over a 12 month period between September 2021 - September 2022.
- Cluster 4: Cluster 4 adverse event data was collected over a 12 month period between September 2021 - September 2022.
- Cluster 5: Cluster 5 adverse event data was collected over a 12 month period between September 2022 - September 2023.
Arm/Group | Cluster 1 | Cluster 2 | Cluster 3 | Cluster 4 | Cluster 5
All-Cause Mortality (participants affected / at risk) | 0/210 | 0/41 | 0/23 | 0/29 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/210 | 0/41 | 0/23 | 0/29 | 0/150
Other Adverse Events (participants affected / at risk) | 0/210 | 0/41 | 0/23 | 0/29 | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03694418/Prot_SAP_002.pdf
  • Informed Consent Form (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03694418/ICF_003.pdf